CLINICAL TRIAL: NCT00116714
Title: Rheumatoid Arthritis Disease Modifying Anti-Rheumatic Drug (DMARD) Intervention and Utilization Study (RADIUS 1)
Brief Title: Rheumatoid Arthritis (DMARD) Intervention and UtilizationStudy
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Collaborators: Immunex Corporation (Industry); Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Other Study IDs: 20021634; 016.0034
Record Dates: First submitted 2005-06-30; First posted 2005-07-01 (Estimated); Last update posted 2011-05-06 (Estimated); Status verified 2011-05

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; RA; DMARD
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Antirheumatic Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Observation
  Interventions: Drug: DMARD

INTERVENTIONS:
Drug: DMARD — All subjects were required to initiate, add or change DMARD therapy at study entry.

SUMMARY:
The Rheumatoid Arthritis DMARD Intervention and Utilization Study (RADIUS 1) is designed to systematically collect and document use patterns, effectiveness, and safety of DMARD treatments currently used in the management of rheumatoid arthritis (RA). It is anticipated that study data may help improve the quality of information upon which clinical decisions are based.

ELIGIBILITY:
Inclusion Criteria:

* Fulfillment of the 1987 American Rheumatism Association criteria for RA
* Currently requiring a new DMARD (change or addition)

Exclusion Criteria:

* Currently enrolled in a clinical trial with treatments or patient visits imposed by a protocol
* Nursing or pregnant women
* Patients with active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with RA according to ACR criteria, and who are starting, adding or changing DMARD therapy, including biologics.
Sampling Method: Non-Probability Sample
Enrollment: 4968 (Actual)
Dates: Start 2001-10; Primary Completion 2007-12 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Gibofsky A, Palmer WR, Keystone EC, Schiff MH, Feng J, McCroskery P, Baumgartner SW, Markenson JA. Rheumatoid arthritis disease-modifying antirheumatic drug intervention and utilization study: safety and etanercept utilization analyses from the RADIUS 1 and RADIUS 2 registries. J Rheumatol. 2011 Jan;38(1):21-8. doi: 10.3899/jrheum.100347. Epub 2010 Oct 15. PMID 20952478
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com